CLINICAL TRIAL: NCT04519671
Title: A Phase IB/IIA Study of Adult Allogeneic Bone Marrow Derived Mesenchymal Stem Cells for the Treatment of Perianal Fistulizing Crohn's Disease
Brief Title: Mesenchymal Stem Cells for the Treatment of Perianal Fistulizing Crohn's Disease
Acronym: PFCD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amy Lightner (Other)
Responsible Party: Sponsor-Investigator, Amy Lightner, Sponsor-Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20-1020
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Perianal Crohn Disease; Perianal Fistula; Crohn Disease
Keywords: perianal fistula; perianal Crohn's disease; mesenchymal stromal cells; mesenchymal stem cells
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mesenchymal Stem Cells (Experimental): Direct injection of adult allogeneic bone marrow derived mesenchymal stem cells, at a dose of 75 million cells into perianal fistula(s) at baseline with a possible repeat injection at 3 months if not completely healed from the first injection.
  Interventions: Drug: Mesenchymal Stem Cells
- Placebo (Placebo Comparator): Direct injection of normal saline. If not completely healed after 6 months, participants will then cross over to the treatment group to receive a direct injection of adult allogeneic bone marrow derived mesenchymal stem cells, at a dose of 75 million cells into perianal fistula(s)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mesenchymal Stem Cells — Direct injection of adult allogeneic bone marrow derived mesenchymal stem cell product, at a dose of 75 million cells into perianal fistula(s)
  Arms: Mesenchymal Stem Cells
Other: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of using adult allogeneic bone marrow derived mesenchymal stem cells (MSCs), to treat people for medically refractory perianal fistulizing Crohn's disease.

DETAILED DESCRIPTION:
Crohn's disease (CD), a chronic transmural inflammatory disease of the gastrointestinal tract, continues to increase in incidence for unknown reasons. According to population based studies, at least 26% of patients with CD will develop perianal fistulas in the first two decades following diagnosis, particularly those with colonic and rectal involvement. These patients experience significant morbidity due to pain, persistent drainage, recurrent perianal sepsis, and ongoing need to access medical care resulting in increased costs and impaired quality of life.

Unfortunately, perianal fistulizing Crohn's disease is notoriously difficult to cure with 37% of patients experiencing refractory disease. As a result, patients cycle through numerous immunosuppressive medications that can have significant side effects, and >90% undergo multiple surgical interventions putting them at risk of incontinence.

The specific rationale for MSCs in perianal Crohn's fistulas is based upon 1) their anti-inflammatory and immunomodulatory properties; 2) several studies reporting the safety and efficacy of MSCs for the treatment of perianal Crohn's fistula; 3) existence of safe manufacturing methods for isolation and expansion of MSCs.

This study will enroll 20 participants that have Crohn's disease with medically and surgically refractory perianal fistulizing disease. Participants enrolled will be those that meet particular criteria for participation in the clinical trial.

Enrolled participants will be randomized to treatment group with adult allogeneic bone marrow derived mesenchymal stem cells, versus placebo in a 3:1 fashion. Participants in the treatment group will have a direct injection of MSCs at a dose of 75 million cells. This will be given as a direct injection in and around the fistula tract. Participants will be evaluated for complete healing at three months. If complete healing has been achieved, participants will continue to be followed for one year. If complete healing has not been achieved at three months, participants will be eligible for a second injection of MSCs at the same dose of 75 million cells. Control participants without complete healing from placebo will cross over at the 6 month visit to receive an injection of MSCs and again three months after this as above, and will be followed for one year after treatment to a total duration of 18 months.

ELIGIBILITY:
Inclusion Criteria

1. Men and Women 18-75 years of age with a diagnosis of Crohn's disease for at least six months duration.
2. Single and Multi-tract Perianal fistula, with or without previous failed surgical repair.
3. Have no contraindications to MR evaluations: e.g. pacemaker or magnetically active metal fragments, claustrophobia
4. Ability to comply with protocol
5. Competent and able to provide written informed consent
6. Concurrent Crohn's-related therapies with stable doses (>2 months) corticosteroids, 5- ASA drugs, immunomodulators, anti-TNF therapy, anti-integrin and anti-interleukin therapies are permitted

Exclusion Criteria

1. Inability to give informed consent.
2. Clinically significant medical conditions within the six months before administration of MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the subject.
3. Specific exclusions:

   1. Hepatitis B or C
   2. HIV
   3. Abnormal AST or ALT at screening(defined as >/= 2x ULN)
4. History of cancer including melanoma (with the exception of localized skin cancers) within one year of screening.
5. History of colorectal cancer within 5 years
6. Investigational drug within one month of treatment
7. Pregnant or breast feeding or trying to become pregnant.
8. Presence of a rectovaginal or perineal body fistula
9. Change in Crohn's immunosuppressive regimen within the 2 months prior to enrollment
10. Uncontrolled intestinal Crohn's disease which will require escalation for medical therapy or surgery within 2 months of enrollment
11. Severe anal canal disease that is stenotic and requires dilation
12. Female participant unwilling to agree to use acceptable contraception methods during participation in study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Treatment related adverse events | Month 6
  Number of participants with treatment related adverse events post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of perianal fistula(s) in the setting of Crohn's disease as assessed by protocol CCF-Stem Cells IBD-001

SECONDARY OUTCOMES:
Complete clinical healing | Month 6, Month 12
  Number of participants with complete clinical healing post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of perianal fistula(s) in the setting of Crohn's disease.
  Complete Healing is defined as:
  Radiographic Healing: MRI with an absence of a fluid collection >2 cm in 3 of 3 dimensions, lack of edema, inflammation or sign of active inflammatory response. A remnant scar of a fistula tract may remain
  Clinical Healing: 100% cessation of drainage on both clinical exam with deep palpation and per patient report and epithelization of the external fistula opening

OTHER OUTCOMES:
Partial clinical healing | Month 6, Month 12
  Number of participants with partial clinical healing post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of perianal fistula(s) in the setting of Crohn's disease
  Partial clinical healing is defined as:
  Radiographic Healing: MRI with an absence of a fluid collection >2 cm in 2 of 3 dimensions, lack of edema, inflammation or sign of active inflammatory response. A remnant scar of a fistula tract may remain
  Clinical healing: Greater than or equal to 50 % cessation of drainage on both clinical exam with deep palpation and per patient report and epithelization of the external fistula opening
Lack of response | Month 6, Month 12
  Number of participants with lack of response post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of perianal fistula(s) in the setting of Crohn's disease
  Lack of response is defined as:
  Radiographic and Clinical healing which does not meet the threshold for Partial Healing
Worsening of disease | Month 6, Month 12
  Number of participants with worsening of disease post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of perianal fistula(s) in the setting of Crohn's disease
  Worsening disease is defined as:
  Radiographic: MRI with a fluid collection >2 cm in 2 of 3 dimensions, edema, inflammation or sign of active inflammatory response. An increased number of tracts may be seen, or increased branching from the primary tract,
  Clinical: Increased drainage per patient report and on clinical exam

CONTACTS AND LOCATIONS:
Overall Officials: Amy Lightner, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kasparek MS, Glatzle J, Temeltcheva T, Mueller MH, Koenigsrainer A, Kreis ME. Long-term quality of life in patients with Crohn's disease and perianal fistulas: influence of fecal diversion. Dis Colon Rectum. 2007 Dec;50(12):2067-74. doi: 10.1007/s10350-007-9006-5. PMID 17680311
- [Background] Sandborn WJ, Fazio VW, Feagan BG, Hanauer SB; American Gastroenterological Association Clinical Practice Committee. AGA technical review on perianal Crohn's disease. Gastroenterology. 2003 Nov;125(5):1508-30. doi: 10.1016/j.gastro.2003.08.025. No abstract available. PMID 14598268
- [Background] Schwartz DA, Loftus EV Jr, Tremaine WJ, Panaccione R, Harmsen WS, Zinsmeister AR, Sandborn WJ. The natural history of fistulizing Crohn's disease in Olmsted County, Minnesota. Gastroenterology. 2002 Apr;122(4):875-80. doi: 10.1053/gast.2002.32362. PMID 11910338
- [Background] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Expanded allogeneic adipose-derived mesenchymal stem cells (Cx601) for complex perianal fistulas in Crohn's disease: a phase 3 randomised, double-blind controlled trial. Lancet. 2016 Sep 24;388(10051):1281-90. doi: 10.1016/S0140-6736(16)31203-X. Epub 2016 Jul 29. PMID 27477896
- [Background] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Diez MC, Tagarro I, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Long-term Efficacy and Safety of Stem Cell Therapy (Cx601) for Complex Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2018 Apr;154(5):1334-1342.e4. doi: 10.1053/j.gastro.2017.12.020. Epub 2017 Dec 24. PMID 29277560
- [Background] Molendijk I, Bonsing BA, Roelofs H, Peeters KC, Wasser MN, Dijkstra G, van der Woude CJ, Duijvestein M, Veenendaal RA, Zwaginga JJ, Verspaget HW, Fibbe WE, van der Meulen-de Jong AE, Hommes DW. Allogeneic Bone Marrow-Derived Mesenchymal Stromal Cells Promote Healing of Refractory Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2015 Oct;149(4):918-27.e6. doi: 10.1053/j.gastro.2015.06.014. Epub 2015 Jun 25. PMID 26116801
- [Background] Molendijk I, van der Meulen-de Jong AE, Verspaget HW, Veenendaal RA, Hommes DW, Bonsing BA, Peeters KCMJ. Standardization of mesenchymal stromal cell therapy for perianal fistulizing Crohn's disease. Eur J Gastroenterol Hepatol. 2018 Oct;30(10):1148-1154. doi: 10.1097/MEG.0000000000001208. PMID 30095479